CLINICAL TRIAL: NCT03822936
Title: Phase II Clinical Study on Resectable or Borderline Resectable Pancreas Adenocarcinoma Preoperative Treatment with Chemotherapy and Carbon Ions Radiation Therapy (hadrontherapy)
Brief Title: Carbon Ions Radiation Therapy for Resectable or Borderline Resectable Pancreas Adenocarcinoma
Acronym: PIOPPO
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was early closed due to low accrual in August 2022.
Sponsor: CNAO National Center of Oncological Hadrontherapy (Other)
Collaborators: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Francesca Valvo, Principal investigator, CNAO National Center of Oncological Hadrontherapy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CNAO 35/2017 C
Record Dates: First submitted 2019-01-25; First posted 2019-01-30 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Cancer of Pancreas; Pancreas Adenocarcinoma; Resectable Pancreatic Cancer
Keywords: carbon ion radiation therapy; exocrine pancreas; pancreas tumour
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Leucovorin; Irinotecan; Fluorouracil; Oxaliplatin; Heavy Ion Radiotherapy

STUDY DESIGN:
Intervention Model Description: The trial enrolls subjects that will receive in order: chemotherapy, carbon ion therapy, followed by surgical resection after 4/6 weeks then adjuvant chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Preoperatory chemoradiation therapy with carbon ions (Experimental): Chemoradiation followed by surgery
  Interventions: Drug: Preoperative chemotherapy; Radiation: Preoperative radiotherapy

INTERVENTIONS:
Drug: Preoperative chemotherapy — Preoperative chemotherapy, carbon ion therapy, surgery
  Other Names: Folinic acid, Irinotecan, fluorouracil, oxaliplatin
Radiation: Preoperative radiotherapy — Preoperative chemotherapy, carbon ion therapy, surgery
  Other Names: Carbon ion therapy

SUMMARY:
Relapses free survival will be evaluated as efficacy of carbon ions radiation therapy released before surgery.

DETAILED DESCRIPTION:
Enrolled subjects will undergo to 3 cycles of Folfirinox before re-evaluation of the lesion. Then, 4D planning and imaging with respiratory gating end rescanning technique will be adopted to calculate the optimal treatment plan to carbon ions radiation therapy: 38.4 Gy[RBE] is the prescribed dose to CTV. 4.8 Gy[RBE]/fraction will be delivered 4 times a week in two weeks. 4/6 weeks after hadrontherapy, after a CT scan with contrast, patient will undergo to a surgery. After 4/6 weeks, Gemcitabine will be administered for 6 cycles.

Secondary endpoints of the trial are overall survival, resectability rate (operable vs borderline operable), acute toxicity within 3 months, 3-6 months, over 6 months.

ELIGIBILITY:
Inclusion Criteria:

* histologic/cytologic diagnosis of exocrine pancreas tumour
* resectable or borderline resectable exocrine pancreatic tumour (according to operability criteria)
* no metastasis from US, CT, PET, MRI or laparotomy
* Karnofsky index >= 70
* stomach and duodenum not infiltrated by tumour
* given informed consent to study procedures
* Hb > 9 g/dL, N> 1500, PLT> 100000
* creatininemia < 1.5 mg/dL; bilirubinemia < 1.5 times upper normal values; albumin > 3 g/dL
* DPD normal activity
* contraception required and breast feeding not permitted

Exclusion Criteria:

* non resectable, locally advanced tumours
* insular cells tumour
* comorbidities excluding abdominal surgery and/or chemo- radiation therapy
* known metastasis
* DPD low activity
* inability to attend study procedures and follow ups
* pregnancy
* previous diagnosis of other tumour with more disadvantageous prognosis then the study object
* metallic biliary stent
* metallic prothesis or any other condition to prevent from target volume individuation and dose calculation
* clinical condition preventing from radiation therapy (i.e. infections in the irradiation area)
* medical and/or psychical condition preventing from radiation therapy
* past radiation therapy on abdomen.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-02-08 (Actual); Primary Completion 2022-08-08 (Actual); Study Completion 2025-02-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival | The local progression free survival will be assessed at 1-year
  The local progression free survival is measured

SECONDARY OUTCOMES:
overall survival | The overall survival of enrolled patients will be assessed at 2-years
  the overall survival of enrolled patients is considered
resectability rate R0 stratified (operable vs not operable) | time of surgery (4-6 weeks after radiotherapy)
  how many surgeries completed according to the procedures and with histopathological margins free from the disease/enrolled patients
Incidence of acute, medium term and late toxicity according to CTCAE v 4.0 grading toxicity | The incidence of acute and medium term toxicity will be assessed up to 90 and 180 post-operative days respectively. The incidence of late toxicity will be assessed through study completion, an average of 1 year.
  Incidence of acute, medium term and late toxicity according to CTCAE v 4.0 grading toxicity
intra and perioperatory complications | The incidence of intra- and perioperatory complications will be assessed up to 30 post-operative days
  intra and perioperatory complications

CONTACTS AND LOCATIONS:
Overall Officials: Francesca Valvo, MD, Principal Investigator — CNAO National Center of Oncological Hadrontherapy
Locations (1):
- CNAO, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barcellini A, Molinelli S, Vanoli A, Vitolo V, Fossati P, Vai A, Pagani A, Inzani F, Pecorilla M, Butturini G, Klersy C, Preda L, Facoetti A, Valvo F, Orlandi E. Preoperative chemo-CIRT in Re/BRe pancreatic cancer: Insights from a multicenter prospective phase II clinical study (NCT03822936). Tumori. 2024 Dec;110(6):470-474. doi: 10.1177/03008916241291341. Epub 2024 Oct 27. PMID 39462835
- [Derived] Vitolo V, Cobianchi L, Brugnatelli S, Barcellini A, Peloso A, Facoetti A, Vanoli A, Delfanti S, Preda L, Molinelli S, Klersy C, Fossati P, Orecchia R, Valvo F. Preoperative chemotherapy and carbon ions therapy for treatment of resectable and borderline resectable pancreatic adenocarcinoma: a prospective, phase II, multicentre, single-arm study. BMC Cancer. 2019 Sep 14;19(1):922. doi: 10.1186/s12885-019-6108-0. PMID 31521134